CLINICAL TRIAL: NCT04362826
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Study to Investigate Efficacy of a Novel Probiotic on the Bacteriome and Mycobiome of Breast Cancer Patients
Brief Title: Study to Investigate Efficacy of a Novel Probiotic on the Bacteriome and Mycobiome of Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CASE13119
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel probiotic (Experimental): Investigational novel probiotic plus normal standard of care for breast cancer.
  Interventions: Biological: Novel probiotic
- Placebo (Placebo Comparator): Placebo plus normal standard of care for breast cancer.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Novel probiotic — Investigational novel probiotic
  Arms: Novel probiotic
Other: Placebo — Placebo for probiotic
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of probiotics on the breast tumor microbiome and gut microbiome in breast cancer. Microorganisms that make up the microbiome (such as viruses, bacteria, and fungi) may have an important role in breast cancer development. Understanding the association of microorganisms with breast cancer may enable new ways to prevent, diagnose, and treat breast cancer.

The probiotic, BIOHM, which is owned and distributed by BIOHM Health LLC, will be used in this study. BIOHM is a food supplement that is believed to balance bacteria and fungi in the body and has received the designation as Generally Recognized as Safe (GRAS) by the Food and Drug Administration (FDA). This study is being done to determine the effectiveness of BIOHM in breast cancer.

DETAILED DESCRIPTION:
This study will investigate the efficacy of the investigational product (a novel probiotic) on altering the microbiome (bacteriomeand mycobiome) and polymicrobial biofilms in the gut of 50 women with breast cancer given the novel probiotic, compared to 50 women with breast cancer given a placebo.

The objectives of this study are to:

1. Determine the efficacy profile of the novel probiotic
2. Analyze bacteriome and mycobiome profiles as well as polymicrobial biofilm composition from breast tissue and stool before and after consumption of the probiotic.
3. Compare quality of life (QoL) of those receiving novel probiotic compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer (invasive ductal carcinoma [IDC] or Invasive Lobular Carcinoma [ILC])
* Minimum breast tumor size of 1.0 cm
* Participants who are of childbearing potential must agree to use a medically approved method of birth control and have a negative pregnancy test result
* BMI between 18.5 to 29.9 kg/m2
* Agree to abstain from consuming unpasteurized bacteria-fermented foods one week prior to baseline visit and throughout the study.
* Agree to not change current dietary habits (apart from avoiding probiotics) and activity/training levels one week prior to screening and during the study.
* Agree to complete all research activities defined in the study
* Participants must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Women who are pregnant, breast feeding, or planning to become pregnant during the trial.
* Use of antibiotics within 5 weeks of randomization.
* History of chronic inflammation or structural abnormality of the digestive tract (e.g., inflammatory bowel disease, duodenal or gastric ulcer intestinal obstruction, or symptomatic cholelithiasis).
* Use of probiotic and/or prebiotic supplements and/or supplemented foods prior to screening and throughout the study.
* Individuals receiving any other investigational agents within 30 days prior to randomization.
* Change in anti-psychotic medication within 3 months prior to randomization.
* Alcohol or drug abuse in the past year.
* Participants with a known allergy to the test material's active or inactive ingredients..

Clinically significant abnormal laboratory results that may negatively impact the participant being involved on the study, at the discretion of the physician.

* Any condition which in the investigators' opinions may adversely affect the participant's ability to complete the study or its measures or which may pose significant risk to the participant.
* Physician feels participation in this trial is not in the subject's best interest.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Beta-D-Glucagon levels | At baseline and at 6 weeks
  Efficacy of the novel probiotic as defined by change in Beta-D-Glucagon levels. This biomarker is well established to measure shifts in the mycobiome
Short-chain fatty acid levels | At baseline and at 6 weeks
  Efficacy of the novel probiotic as defined by change in short-chain fatty acid levels. This biomarker is well established to measure shifts in the bacteriome
Free amino acid levels | At baseline and at 6 weeks
  Efficacy of the novel probiotic as defined by change in free amino acid levels. This biomarker is well established to measure shifts in the bacteriome

SECONDARY OUTCOMES:
Alpha and beta biodiversity of gut microbiome and mycobiome | At baseline and at 6 weeks
  Gut microbiome and polymicrobioal biofilm composition analyzed through bacteriome in stool as measured by alpha and beta biodiversity
Differential abundances of gut microbiome and mycobiome | At baseline and at 6 weeks
  Gut microbiome and polymicrobioal biofilm composition analyzed through bacteriome in stool as measured by differential abundances
Polymicrobial biofilm composition of gut microbiome and mycobiome | At baseline and at 6 weeks
  Gut microbiome and polymicrobioal biofilm composition analyzed through bacteriome in stool as measured by polymicrobioal biofilm composition
Alpha and beta biodiversity of breast microbiome and mycobiome | At baseline and at 6 weeks
  Gut microbiome and polymicrobioal biofilm composition analyzed through bacteriome in breast tissue as measured by alpha and beta biodiversity
Differential abundances of breast microbiome and mycobiome | At baseline and at 6 weeks
  Gut microbiome and polymicrobioal biofilm composition analyzed through bacteriome in breast tissue as measured by differential abundances
Polymicrobial biofilm composition of breast microbiome and mycobiome | At baseline and at 6 weeks
  Gut microbiome and polymicrobioal biofilm composition analyzed through bacteriome in breast tissue as measured by polymicrobioal biofilm composition
QoL via standardized European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 | At baseline and at 6 weeks
  Quality of life (QoL) via EORTC QLQ C-30 will be converted into dimensions, which evaluate the quality of life associated with health. Dimensions are expected to range 0-100, with high scores referring to higher responses (QoL, symptoms) and are described by the arithmetic mean and standard deviation. Mann-Whitney U test will be utilized to compare the dimensions between each of the 2 groups (probiotic vs placebo groups). For testing the statistical significance of the change in dimensions before and after treatment (within probiotic arm; within placebo arm), the Wilcoxon signed rank test will be used. P<0.05 will be considered statistically significant.
QoL via EORTC QLQ-BR23 | At baseline and at 6 weeks
  EORTC QLQ-BR23 will be converted into dimensions, which evaluate the quality of life associated with health. Dimensions are expected to range 0-100 with high scores referring to higher responses (QoL, symptoms) and are described by the arithmetic mean and standard deviation. Mann-Whitney U test will be utilized to compare the dimensions between each of the 2 groups (probiotic vs placebo groups). For testing the statistical significance of the change in dimensions before and after treatment (within probiotic arm; within placebo arm), the Wilcoxon signed rank test will be used. P<0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Zahraa Al-Hilli, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication
Supporting Information: Study Protocol, SAP, ICF